CLINICAL TRIAL: NCT01154647
Title: Unraveling Impaired Pain Inhibition in Patients With Rheumatoid Arthritis and Central Sensitivity Syndromes: a Series of Experiments Targeting Brain Neurotransmission
Brief Title: Pain Inhibition in Patients With Rheumatoid Arthritis and Central Sensitivity Syndromes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Research Foundation Flanders (Other); Universiteit Antwerpen (Other); University Hospital, Antwerp (Other); Artesis University College, Antwerp (Other)
Responsible Party: Meeus, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: EudraCT 2010-020498-17
Record Dates: First submitted 2010-06-28; First posted 2010-07-01 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2010-04

CONDITIONS: Fatigue Syndrome, Chronic; Fibromyalgia; Arthritis, Rheumatoid
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fibromyalgia; Arthritis, Rheumatoid | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- selective serotonin reuptake inhibitor (Experimental): intravenous, acute, 20mg/ml
  Interventions: Drug: citalopram
- 1 ml 0.9 % NaCl (Placebo Comparator)
  Interventions: Drug: 1 ml 0.9 % NaCl

INTERVENTIONS:
Drug: citalopram — intravenous
  Arms: selective serotonin reuptake inhibitor
Drug: 1 ml 0.9 % NaCl — intravenous
  Arms: 1 ml 0.9 % NaCl

SUMMARY:
Both patients with peripheral structural pathologies, like rheumatoid arthritis (RA)-patients, or patients with central sensitivity syndromes (CSS) suffer chronic pain. CSS are characterized by an increased responsiveness of central pain neurons. An impaired endogenous pain inhibition is already demonstrated in CSS. In the present study the investigators want to evaluate the efficacy of pain inhibition in response to physical stressors and whether the efficacy is opioid-mediated in two chronic pain populations (RA & CCS) compared to controls.

Therefore a triple-blinded randomized controlled trial (RCT) with cross-over design will be performed. The efficacy of wind-up of pain and spatial summation of pain is evaluated before and after a submaximal exercise, while the experimental group receives a selective serotonin reuptake inhibitor. Participants are 20 RA-patients and 20 CSS-patients, more specific patients with fibromyalgia and chronic fatigue syndrome, and 30 healthy controls. This way, the investigators analyze how pain inhibition reacts on different types of physical stressors in different pain patients and if pain inhibition is opioid-mediated.

ELIGIBILITY:
Inclusion Criteria:

* Each study participant should be aged between 18 and 65 years. All three groups will be comparable for age, gender, education level and socioeconomic status; both patient groups will be comparable for illness duration.
* The Central Sensitivity Syndrome (CSS) group will comply with the diagnostic criteria for Fibromyalgia (FM) as defined by the American College of Rheumatology and the Centre of Disease Control criteria for Chronic Fatigue Syndrome (CFS).
* At the time of study participation, healthy control subjects cannot suffer any pain complaints. Sedentary is defined as a sedentary job and < 3 h moderate physical activity/week. Moderate physical activity is defined as activity demanding at least the threefold of the energy spent passively.
* Patients have to be able to cycle on a bicycle ergometer.

Exclusion Criteria:

* In order to preclude confounding factors, participants cannot be pregnant (pregnancy test) or until 1 year postnatal and will be asked to stop medication two weeks prior to study participation, not to undertake physical exertion, and to refrain from consuming caffeine, alcohol or nicotine on the day of the experiment. For ethical reasons, Rheumatoid arthritis(RA)-patients are able to take non-opioid pain medication as described in the 1st step of the World Health Organization analgesic ladder (Non-Steroidal Anti-Inflammatory Drugs and paracetamol).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Pain rates according to a visual analogue scale upon repeated pulses at pressure pain detection threshold intensity | 5 minutes before and after exercise
  Temporal summation is elicited with 10 pulses of the algometer at pressure pain detection threshold intensity on the dorsal surface of the right hand middle finger midway between the first and the second digital joints, and at the trapezius. Subjects are instructed to rate the pain level of the 1st, 5th and 10th pulse according to a visual analogue scale (VAS).
  To assess spatial summation an occlusion cuff inflated to a painful intensity and maintained at that level while repeated algometer pulses are administered and pain ratings are recorded again.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

REFERENCES:
- [Derived] Meeus M, Hermans L, Ickmans K, Struyf F, Van Cauwenbergh D, Bronckaerts L, De Clerck LS, Moorken G, Hans G, Grosemans S, Nijs J. Endogenous pain modulation in response to exercise in patients with rheumatoid arthritis, patients with chronic fatigue syndrome and comorbid fibromyalgia, and healthy controls: a double-blind randomized controlled trial. Pain Pract. 2015 Feb;15(2):98-106. doi: 10.1111/papr.12181. Epub 2014 Feb 17. PMID 24528544